CLINICAL TRIAL: NCT00792298
Title: A Phase IIb, Multicenter, Randomized, Double-Blind Placebo-Controlled, 2-period Adaptive Crossover Polysomnography Study to Evaluate Safety and Efficacy of MK-4305 in Patients With Primary Insomnia
Brief Title: Phase IIB 2-Period Crossover Polysomnography Study in Participants With Primary Insomnia (MK-4305-006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4305-006; 2008_583 (Other: Merck Registration Number)
Record Dates: First submitted 2008-11-10; First posted 2008-11-17 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- Suvorexant 10 mg → Placebo (Experimental): After an ~1- to 2-week single-blind placebo run-in period, participants received 10 mg suvorexant daily prior to bedtime for 4 weeks during Treatment Period 1, followed by a 1-week single-blind placebo washout period, followed by dose-matched placebo to suvorexant daily prior to bedtime during Treatment Period 2.
  Interventions: Drug: Suvorexant; Drug: Dose-matched Placebo to Suvorexant
- Placebo → Suvorexant 10 mg (Experimental): After an ~1- to 2-week single-blind placebo run-in period, participants received dose-matched placebo to suvorexant daily prior to bedtime for 4 weeks during Treatment Period 1, followed by a 1-week single-blind placebo washout period, followed by 10 mg suvorexant daily prior to bedtime during Treatment Period 2.
  Interventions: Drug: Suvorexant; Drug: Dose-matched Placebo to Suvorexant
- Suvorexant 20 mg → Placebo (Experimental): After an ~1- to 2-week single-blind placebo run-in period, participants received 20 mg suvorexant daily prior to bedtime for 4 weeks during Treatment Period 1, followed by a 1-week single-blind placebo washout period, followed by dose-matched placebo to suvorexant daily prior to bedtime during Treatment Period 2.
  Interventions: Drug: Suvorexant; Drug: Dose-matched Placebo to Suvorexant
- Placebo → Suvorexant 20 mg (Experimental): After an ~1- to 2-week single-blind placebo run-in period, participants received dose-matched placebo to suvorexant daily prior to bedtime for 4 weeks during Treatment Period 1, followed by a 1-week single-blind placebo washout period, followed by 20 mg suvorexant daily prior to bedtime during Treatment Period 2.
  Interventions: Drug: Suvorexant; Drug: Dose-matched Placebo to Suvorexant
- Suvorexant 40 mg → Placebo (Experimental): After an ~1- to 2-week single-blind placebo run-in period, participants received 40 mg suvorexant daily prior to bedtime for 4 weeks during Treatment Period 1, followed by a 1-week single-blind placebo washout period, followed by dose-matched placebo to suvorexant daily prior to bedtime during Treatment Period 2.
  Interventions: Drug: Suvorexant; Drug: Dose-matched Placebo to Suvorexant
- Placebo → Suvorexant 40 mg (Experimental): After an ~1- to 2-week single-blind placebo run-in period, participants received dose-matched placebo to suvorexant daily prior to bedtime for 4 weeks during Treatment Period 1, followed by a 1-week single-blind placebo washout period, followed by 40 mg suvorexant daily prior to bedtime during Treatment Period 2.
  Interventions: Drug: Suvorexant; Drug: Dose-matched Placebo to Suvorexant
- Suvorexant 80 mg → Placebo (Experimental): After an ~1- to 2-week single-blind placebo run-in period, participants received 80 mg suvorexant daily prior to bedtime for 4 weeks during Treatment Period 1, followed by a 1-week single-blind placebo washout period, followed by dose-matched placebo to suvorexant daily prior to bedtime during Treatment Period 2.
  Interventions: Drug: Suvorexant; Drug: Dose-matched Placebo to Suvorexant
- Placebo → Suvorexant 80 mg (Experimental): After an ~1- to 2-week single-blind placebo run-in period, participants received dose-matched placebo to suvorexant daily prior to bedtime for 4 weeks during Treatment Period 1, followed by a 1-week single-blind placebo washout period, followed by 80 mg suvorexant daily prior to bedtime during Treatment Period 2.
  Interventions: Drug: Suvorexant; Drug: Dose-matched Placebo to Suvorexant

INTERVENTIONS:
Drug: Suvorexant — oral tablet taken before bedtime
  Other Names: MK-4305
Drug: Dose-matched Placebo to Suvorexant — Dose-matched placebo to suvorexant taken before bedtime (oral tablet)

SUMMARY:
A cross-over, polysomnography study to test the safety, tolerability and effectiveness of different doses of suvorexant (MK-4305) in the treatment of patients with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of Primary Insomnia based on sleep history and the investigator's judgment
* Must be willing to stay overnight at a sleep laboratory
* Must be willing to stay in bed for at least 8 hours each night while at the sleep laboratory
* Regular bedtime is between 9 PM and 12 AM (midnight)

Exclusion Criteria:

* Breast feeding, pregnant or planning to become pregnant during the study
* Within the past 6 months before starting the study you have a history of significant cardiovascular disorder such as unstable angina, congestive heart - failure or acute coronary syndrome
* Currently participating or have participated in a study with an investigational compound or device within the last 30 days
* Has traveled across 3 or more time zones in the last 2 weeks or plans on traveling across 3 or more time zones at any time during the study
* Has done shift work within the past 2 weeks
* Has donated blood products within the last 8 weeks
* Has difficulty sleeping due to a medical condition

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2008-11-05 (Actual); Primary Completion 2009-12-26 (Actual); Study Completion 2009-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Herring WJ, Snyder E, Budd K, Hutzelmann J, Snavely D, Liu K, Lines C, Roth T, Michelson D. Orexin receptor antagonism for treatment of insomnia: a randomized clinical trial of suvorexant. Neurology. 2012 Dec 4;79(23):2265-74. doi: 10.1212/WNL.0b013e31827688ee. Epub 2012 Nov 28. PMID 23197752
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=4305-006&kw=4305-006&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Suvorexant 10 mg → Placebo | Placebo → Suvorexant 10 mg | Suvorexant 20 mg → Placebo | Placebo → Suvorexant 20 mg | Suvorexant 40 mg → Placebo | Placebo → Suvorexant 40 mg | Suvorexant 80 mg → Placebo | Placebo → Suvorexant 80 mg
Started | 31 | 32 | 33 | 32 | 32 | 32 | 31 | 31
Completed | 30 | 31 | 31 | 28 | 32 | 29 | 27 | 30
Not Completed | 1 | 1 | 2 | 4 | 0 | 3 | 4 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout
Arm/Group | Suvorexant 10 mg → Placebo | Placebo → Suvorexant 10 mg | Suvorexant 20 mg → Placebo | Placebo → Suvorexant 20 mg | Suvorexant 40 mg → Placebo | Placebo → Suvorexant 40 mg | Suvorexant 80 mg → Placebo | Placebo → Suvorexant 80 mg
Started | 30 | 31 | 32 (1 participant discontinued therapy during Period 1 but entered the Washout as allowed per protocol) | 28 | 32 | 29 | 29 (2 participants discontinued therapy during Period 1 but entered the Washout as allowed per protocol) | 30
Completed | 30 | 31 | 31 | 28 | 32 | 27 | 29 | 30
Not Completed | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Period: Treatment Period 2
Arm/Group | Suvorexant 10 mg → Placebo | Placebo → Suvorexant 10 mg | Suvorexant 20 mg → Placebo | Placebo → Suvorexant 20 mg | Suvorexant 40 mg → Placebo | Placebo → Suvorexant 40 mg | Suvorexant 80 mg → Placebo | Placebo → Suvorexant 80 mg
Started | 30 | 31 | 31 | 28 | 32 | 27 | 29 | 30
Completed | 29 | 30 | 30 | 26 | 30 | 27 | 28 | 28
Not Completed | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Treated Participants: All randomized participants who received at least one dose of study treatment.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148
  Male | 106

OUTCOME MEASURES:

1. Primary Outcome: LS Mean Sleep Efficiency (SE) During Periods 1 and 2
Description: SE was defined as total sleep time (TST) in minutes divided by time in bed (measured from lights off to lights on; fixed at 8 hours on each Polysomnography [PSG] night) in minutes, multiplied by 100, where TST is defined as the total time (minutes) in Stages 1, 2, 3, 4 and Rapid Eye Movement (REM). SE= (total sleep time/time in bed) x 100
Time Frame: Night 1 and end of Week 4
Population: Full Analysis Set (FAS) population; subset of all randomized participants who received at least one dose of study medication and had any post-randomization efficacy assessment data. The FAS population may have varied across endpoints due to the degree of missing data for each endpoint.
Measure: Least Squares Mean (Standard Error); unit: percent of time in bed
Groups:
- Placebo: Participants received dose-matched placebo to suvorexant daily prior to bedtime over a 4-week treatment period.
- Suvorexant 10 mg: Participants received 10 mg suvorexant daily prior to bedtime over a 4-week treatment period.
- Suvorexant 20 mg: Participants received 20 mg suvorexant daily prior to bedtime over a 4-week treatment period.
- Suvorexant 40 mg: Participants received 40 mg suvorexant daily prior to bedtime over a 4-week treatment period.
- Suvorexant 80 mg: Participants received 80 mg suvorexant daily prior to bedtime over a 4-week treatment period.
Arm/Group | Placebo | Suvorexant 10 mg | Suvorexant 20 mg | Suvorexant 40 mg | Suvorexant 80 mg
Number analyzed (Participants) | 249 | 62 | 61 | 59 | 61
percent of time in bed
  Night 1 (n=249, 62, 61, 59, 61) | 75.8 (0.93) [74.0 to 77.6] | 81.0 (1.75) [77.6 to 84.5] | 83.4 (1.75) [79.9 to 86.8] | 86.6 (1.77) [83.1 to 90.1] | 88.7 (1.77) [85.2 to 92.2]
  Week 4 (n=232, 59, 57, 57, 55) | 76.6 (0.94) [74.8 to 78.5] | 81.3 (1.66) [78.0 to 84.6] | 87.0 (1.68) [83.7 to 90.3] | 84.4 (1.68) [81.1 to 87.7] | 84.2 (1.70) [80.9 to 87.6]
Statistical Analysis 1: Comparison: Placebo vs Suvorexant 80 mg; A fixed sequential testing procedure assessed statistical significance, beginning with the highest dose. The comparison of suvorexant vs placebo had to be significant at α=0.05 at both Night 1 and Week 4 in order to assess statistical significance of the comparison of suvorexant vs placebo for the next highest dose. If a non-significant result was observed at either time point, the differences between suvorexant and placebo for SE was considered nonsignificant for this and all lower doses; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = 12.9, 95% CI 2-sided [9.5 to 16.3]
Statistical Analysis 2: Comparison: Placebo vs Suvorexant 80 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Week 4 = 7.6, 95% CI 2-sided [4.4 to 10.9]
Statistical Analysis 3: Comparison: Placebo vs Suvorexant 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = 10.8, 95% CI 2-sided [7.4 to 14.2]
Statistical Analysis 4: Comparison: Placebo vs Suvorexant 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Week 4 = 7.8, 95% CI 2-sided [4.6 to 10.9]
Statistical Analysis 5: Comparison: Placebo vs Suvorexant 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = 7.6, 95% CI 2-sided [4.2 to 11.0]
Statistical Analysis 6: Comparison: Placebo vs Suvorexant 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Week 4 = 10.4, 95% CI 2-sided [7.2 to 13.6]
Statistical Analysis 7: Comparison: Placebo vs Suvorexant 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; LS Mean Difference: Night 1 = 5.2, 95% CI 2-sided [1.9 to 8.6]
Statistical Analysis 8: Comparison: Placebo vs Suvorexant 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; LS Mean Difference: Week 4 = 4.7, 95% CI 2-sided [1.6 to 7.8]

2. Secondary Outcome: LS Mean Wake After Persistent Sleep Onset (WASO) During Periods 1 and 2
Description: WASO was defined as the duration of wakefulness measured in minutes (any epoch of Stage 0) from persistent sleep onset (first epoch of the first twenty consecutive epochs of non-wake) to lights on.
Time Frame: Night 1 and end of Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | Suvorexant 10 mg | Suvorexant 20 mg | Suvorexant 40 mg | Suvorexant 80 mg
Number analyzed (Participants) | 249 | 62 | 61 | 59 | 61
minutes
  Night 1 (n=249, 62, 61, 59, 61) | 72.4 (3.38) [65.8 to 79.1] | 51.3 (6.40) | 47.7 (6.41) | 38.5 (6.47) | 35.6 (6.46)
  Week 4 (n=232, 59, 57, 57, 55) | 76.7 (3.60) [69.6 to 83.7] | 55.2 (6.65) | 48.6 (6.75) | 43.4 (6.77) | 47.8 (6.84)
Statistical Analysis 1: Comparison: Placebo vs Suvorexant 80 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = -36.8, 95% CI 2-sided [-49.4 to -24.3]
Statistical Analysis 2: Comparison: Placebo vs Suvorexant 80 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Week 4 = -28.9, 95% CI 2-sided [-42.1 to -15.7]
Statistical Analysis 3: Comparison: Placebo vs Suvorexant 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = -33.9, 95% CI 2-sided [-46.4 to -21.5]
Statistical Analysis 4: Comparison: Placebo vs Suvorexant 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Week 4 = -33.2, 95% CI 2-sided [-46.3 to -20.2]
Statistical Analysis 5: Comparison: Placebo vs Suvorexant 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = -24.7, 95% CI 2-sided [-37.1 to -12.3]
Statistical Analysis 6: Comparison: Placebo vs Suvorexant 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Week 4 = -28.1, 95% CI 2-sided [-41.0 to -15.1]
Statistical Analysis 7: Comparison: Placebo vs Suvorexant 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = -21.2, 95% CI 2-sided [-33.5 to -8.8]
Statistical Analysis 8: Comparison: Placebo vs Suvorexant 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; LS Mean Difference: Week 4 = -21.4, 95% CI 2-sided [-34.2 to -8.7]

3. Secondary Outcome: LS Mean Latency to the Onset of Persistent Sleep (LPS) During Periods 1 and 2
Description: LPS is defined as the duration of time measured in minutes from lights off to persistent sleep onset.
Time Frame: Night 1 and end of Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | Suvorexant 10 mg | Suvorexant 20 mg | Suvorexant 40 mg | Suvorexant 80 mg
Number analyzed (Participants) | 249 | 62 | 61 | 59 | 61
minutes
  Night 1 (n=249, 62, 61, 59, 61) | 49.8 (2.91) | 46.4 (6.08) | 40.4 (6.08) | 26.7 (6.13) | 24.4 (6.13)
  Week 4 (n=232, 59, 57, 57, 55) | 41.7 (2.75) | 39.4 (5.12) | 19.4 (5.17) | 37.9 (5.19) | 32.2 (5.28)
Statistical Analysis 1: Comparison: Placebo vs Suvorexant 80 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = -25.4, 95% CI 2-sided [-37.7 to -13.1]
Statistical Analysis 2: Comparison: Placebo vs Suvorexant 80 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.068, Mixed Models Analysis; LS Mean Difference: Week 4 = -9.5, 95% CI 2-sided [-19.7 to 0.7]
Statistical Analysis 3: Comparison: Placebo vs Suvorexant 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = -23.1, 95% CI 2-sided [-35.3 to -10.9]
Statistical Analysis 4: Comparison: Placebo vs Suvorexant 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.459, Mixed Models Analysis; LS Mean Difference: Week 4 = -3.8, 95% CI 2-sided [-13.8 to 6.3]
Statistical Analysis 5: Comparison: Placebo vs Suvorexant 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.130, Mixed Models Analysis; LS Mean Difference: Night 1 = -9.4, 95% CI 2-sided [-21.5 to 2.8]
Statistical Analysis 6: Comparison: Placebo vs Suvorexant 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Week 4 = -22.3, 95% CI 2-sided [-32.3 to -12.3]
Statistical Analysis 7: Comparison: Placebo vs Suvorexant 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.577, Mixed Models Analysis; LS Mean Difference: Night 1 = -3.4, 95% CI 2-sided [-15.6 to 8.7]
Statistical Analysis 8: Comparison: Placebo vs Suvorexant 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.644, Mixed Models Analysis; LS Mean Difference: Week 4 = -2.3, 95% CI 2-sided [-12.2 to 7.5]

4. Post Hoc Outcome: LS Mean Latency to the Onset of Persistent Sleep (LPS) During Period 1 (To Exclude Carryover Effect)
Description: LPS is defined as the duration of time measured in minutes from lights off to persistent sleep onset. In order to evaluate the efficacy of suvorexant on LPS excluding the influence of a carryover effect from Period 1 to Period 2, an ad hoc analysis of LPS restricted to Period 1 data was also performed.
Time Frame: Night 1 (Period 1 only) and end of Week 4 (Period 1 only)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Groups:
- Placebo: Participants received dose-matched placebo to suvorexant daily prior to bedtime over 4 weeks in Treatment Period 1.
- Suvorexant 10 mg: Participants received 10 mg suvorexant daily prior to bedtime over 4 weeks in Treatment Period 1.
- Suvorexant 20 mg: Participants received 20 mg suvorexant daily prior to bedtime over 4 weeks in Treatment Period 1.
- Suvorexant 40 mg: Participants received 40 mg suvorexant daily prior to bedtime over 4 weeks in Treatment Period 1.
- Suvorexant 80 mg: Participants received 80 mg suvorexant daily prior to bedtime over 4 weeks in Treatment Period 1.
Arm/Group | Placebo | Suvorexant 10 mg | Suvorexant 20 mg | Suvorexant 40 mg | Suvorexant 80 mg
Number analyzed (Participants) | 127 | 31 | 33 | 32 | 31
minutes
  Night 1 (n=127, 31, 33, 32, 31) | 57.0 (4.29) | 38.0 (7.67) | 39.6 (7.41) | 26.0 (7.56) | 34.7 (7.67)
  Week 4 (n=116, 29, 31, 30, 28) | 52.4 (4.43) | 32.2 (7.97) | 27.7 (7.71) | 36.6 (7.88) | 32.8 (8.07)
Statistical Analysis 1: Comparison: Placebo vs Suvorexant 80 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; LS Mean Difference: Night 1 = -22.3, 95% CI 2-sided [-38.3 to -6.2]
Statistical Analysis 2: Comparison: Placebo vs Suvorexant 80 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis; LS Mean Difference: Week 4 = -19.6, 95% CI 2-sided [-36.6 to -2.6]
Statistical Analysis 3: Comparison: Placebo vs Suvorexant 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference: Night 1 = -31.0, 95% CI 2-sided [-46.9 to -15.2]
Statistical Analysis 4: Comparison: Placebo vs Suvorexant 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.063, Mixed Models Analysis; LS Mean Difference: Week 4 = -15.7, 95% CI 2-sided [-32.3 to 0.8]
Statistical Analysis 5: Comparison: Placebo vs Suvorexant 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis; LS Mean Difference: Night 1 = -17.4, 95% CI 2-sided [-33.1 to -1.7]
Statistical Analysis 6: Comparison: Placebo vs Suvorexant 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; LS Mean Difference: Week 4 = -24.6, 95% CI 2-sided [-41.0 to -8.3]
Statistical Analysis 7: Comparison: Placebo vs Suvorexant 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis; LS Mean Difference: Night 1 = -19.1, 95% CI 2-sided [-35.1 to -3.0]
Statistical Analysis 8: Comparison: Placebo vs Suvorexant 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis; LS Mean Difference: Week 4 = -20.2, 95% CI 2-sided [-37.0 to -3.4]

ADVERSE EVENTS:
Arm/Group | Placebo | Suvorexant 10 mg | Suvorexant 20 mg | Suvorexant 40 mg | Suvorexant 80 mg
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/62 | 0/61 | 0/59 | 0/61
Other Adverse Events (participants affected / at risk) | 9/249 | 1/62 | 4/61 | 11/59 | 11/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=249) | Suvorexant 10 mg (N=62) | Suvorexant 20 mg (N=61) | Suvorexant 40 mg (N=59) | Suvorexant 80 mg (N=61)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 7 (7) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.